CLINICAL TRIAL: NCT04022187
Title: Assessment of the Excitability of Spinal Motoneurons Using Stimulus-response Curves of the Bulbocavernosus Reflex
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon Hospital, Pierre and Marie Curie University
Other Study IDs: PGRC 001 GREEN
Record Dates: First submitted 2019-07-13; First posted 2019-07-17 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Spasticity, Muscle
Keywords: Bulbocavernosus reflex; Spasticity assessment; Motoneurone excitability; Stimulus-response curves
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bulbocavernosus reflex assessment: Patients over 18 years old, consulting in neuro-urology department for urinary, anorectal or genito-sexual disorders.
  Interventions: Other: Observational study : no intervention

INTERVENTIONS:
Other: Observational study : no intervention — Observational study : no intervention, only exporting data

SUMMARY:
Spasticity is commonly observed in neurological conditions such as Multiple Sclerosis and spinal cord injury. "Peripheral" spasticity, concerning in particular the striated muscles of the limbs is nowadays well known and studied with clinical scales (Ashworth, Taridieu...) or even electrophysiological methods (H-reflex, T-reflex...). However, this spasticity can also affect the perineal muscles and more generally the pelvic muscles. However, there is to date no validated and standardized method for evaluating this pelvi-perineal spasticity.

The aim of the study will be to assess the spinal motoneurons excitability by using the stimulus-response curves of the bulbocavernosus reflex.

DETAILED DESCRIPTION:
Spasticity defined by Lance in 1980 is "a motor disorder characterized by a velocity dependent increase in the tonic stretch reflexes (muscle tone) with exaggerated tendon jerks, resulting from hyperexcitability of the stretch reflexes as one component of the upper motor neuron syndrome". The occurrence of spasticity, which is common in neurology when the pyramidal tract is affected, is commonly observed in the "peripheral" striated muscles. However, spasticity also concerns the perineal musculature, with "the exaggeration of the stretching reflex of the muscles accessible to pelvic touches". Although there are measurement scales commonly used in clinical practice, such as the Ashworth and Tardieu scales, or electrophysiological instrumental techniques (H reflex , T reflex), there is actually no objective and standardized measurement technique for pelvic spasticity. An interesting tool could be the bulbocavernosus reflex (BCR) which is a polysynaptic reflex with sacral integration. In addition to its diagnostic and topographical value due to its sacral integration, BCR could testify, by its modulation, to the control of the alpha motor neuron pool. It could therefore allow to assess motoneuronal excitability, whose increase may lead in central patients with supra-connal lesions (spinal cord injuries (SCI), multiple sclerosis (MS)), to a release of sacral automatism with exacerbation of reflex responses whether bladder (detrusor overactivity), sphincter (detrusor-sphincter dysynergia) or rectal (rectal overactivity).

The aim of the study will be to assess the sacral spinal motor neuron excitability using the stimulus-response curves of the BCR.

The investigators will conduct a prospective monocentric observational study in a specialized neuro-urology department. The main objective of this study will be to evaluate the spinal motoneuron excitability according to the degree of bladder repletion by modelling recruitment slopes (stimulus-response curves) of the BCR.

First of all, the investigators will assess the feasibility of conducting an analysis of BCR stimulus-response curves during a perineal electrophysiological exploration performed in a diagnostic context in patients referred for urinary, anorectal or genito-sexual disorders. BCR will be recorded after electrical stimulation of the dorsal nerve of the penis or the dorsal nerve of the clitoris, using a concentric needle electrode inserted into the left and then right bulbcavernous muscle. Stimulations will be performed at progressively increasing intensities and each response will be recorded. Acquisition will be performed using a Dantec™ Keypoint® G4 EMG device, Natus®. The initial stimulation intensity will be at the motor threshold, i.e. the degree of stimulation that determines a stable latent motor response and will then be increased by 10 to 10 mA to obtain the following 4 reflex responses. Once the acquisition will be completed, the curves will be analyzed allowing the analysis of the area under the curve (AUC) and the construction of the stimulus-response curves.

In a second step, the investigators will evaluate the possibility of modelling these stimulus-response curves after EMG recording using pre-gelled disposable surface electrodes placed on the external anal sphincter (EAS) during a cystometry performed in patients consulting for urinary disorders. The stimulation technique will be identical as described previously. Finally, the modulation of spinal motoneurons excitability according to the degree of bladder filling will be assessed by modelling the BCR stimulus-response curves, before and during a cystometry.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old minimum
* Subjects with spinal cord injury or multiple sclerosis, requiring an electrophysiological and urodynamic explorations in our neuro-urology specialized department, with a strictly supra-sacral central neurological condition.
* Subjects with stress urinary incontinence (SUI) requiring perineal explorations including a cystometry and a perineal EMG.

Exclusion Criteria:

* Subjects with peripheral neurological impairment (cauda equina syndrome, medullary cone syndrome, advanced diabetes)
* Subjects who received a treatment by injection of intra-detrusorian botulinum toxin in the last 6 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who will be referred to our specialized neuro-urology service for electrophysiological and urodynamic explorations
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Variation of the recruitment slope according to the degree of bladder repletion | 1 day
  For each patient, an assessment of spinal motoneuron excitability by using the area under the motor response curve of the bulbocavernous reflex will be performed before starting the cystometry (empty bladder) and during urgent urination needs (also during the cystometry) to determine an alpha angle of the recruitment curve. The primary outcome is the variation in this alpha coefficient.

SECONDARY OUTCOMES:
Comparison of the variation of recruitment slope according to the bladder repletion : (empty bladder - B1) versus (B1-B3) variation | 1 day
Influence of neurological disease on spinal motoneuron excitability | 1 day
  comparison of the variation of the recruitment slope observed in neurological subjects versus non-neurological subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PHD, Principal Investigator — Sorbonne Université, GRC 001, GREEN, AP-HP, Hôpital Tenon, Paris, France
Locations (1):
- Department of neuro-urology, hôpital Tenon, Paris, France